CLINICAL TRIAL: NCT00389324
Title: An Open-Label Single-Sequence, Crossover Trial to Evaluate the Pharmacokinetics and Safety of Subcutaneous Gamunex® 10% (Immune Globulin Intravenous [Human], 10% Caprylate/Chromatography Purified) in Subjects With Primary Immunodeficiency
Brief Title: A Trial of the Pharmacokinetics, Safety, and Tolerability of Subcutaneous Gamunex® in Primary Immunodeficiency
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Grifols Therapeutics LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 060001
Record Dates: First submitted 2006-10-17; First posted 2006-10-18 (Estimated); Results first posted 2012-12-18 (Estimated); Last update posted 2015-04-20 (Estimated); Status verified 2015-03

CONDITIONS: Immunologic Deficiency Syndrome
Keywords: Primary immune deficiency
MeSH Terms: conditions — Immunologic Deficiency Syndromes; Primary Immunodeficiency Diseases | interventions — Immunoglobulins, Intravenous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Immune Globulin Intravenous (Human) (Experimental): Immune Globulin Intravenous (Human), 10%, Caprylate/Chromatography Purified
  Interventions: Biological: Immune Globulin Intravenous (Human)

INTERVENTIONS:
Biological: Immune Globulin Intravenous (Human) — This trial was an open-label, single-sequence, study. The enrolled subjects received IGIV-C via two routes of administration (IV for 4 -5 weeks and SC for 24 weeks) in order to compare the PK variables, safety and tolerability of SC administration of IGIV-C. Certain subjects required IV IGIV-C dosing during a Run-in Phase (3 - 4 months) for steady-state conditions prior to the IV phase. Subjects received two IV infusions of IGIV (between 200 - 600 mg based on the subject's previous IgG dosing regimen, 3 to 4 weeks apart) until a steady-state was reached at which time PK profiling was performed. Subjects began weekly SC administration (1.37 times the weekly equivalency of each subject's monthly IV dose) 1 week following last IV dose and followed for a period of six months.
  Other Names: Gamunex; Gaminex; Immune globulin intravenous (Human)(IGIV); BAY 41-1000; TAL-05-00004; IGIV-C; IVIG; IGIVnex; NDC-13353-645-71; NDC-13353-646-24; NDC-13353-645-12; NDC-13353-645-15; NDC-13353-645-2

SUMMARY:
This study will compare the blood level of Gamunex in patients. Patients will take it as an injection under the skin or in a vein. The study will compare how safe and tolerable the two methods are in the patients. The patients in this study have a defect in their immune system from a genetic cause.

DETAILED DESCRIPTION:
This is an open-label, single-sequence, multi-center trial with subjects previously diagnosed with primary immune deficiency. Subjects will be on IGIV until a steady state is reached at which time PK profiling during the IV phase will occur. Subjects will begin SC administration 1 week following last IV dose and followed for a period of six months. PK profiling in SC phase will occur when subject reaches approximate steady-state on SC administration.

ELIGIBILITY:
Inclusion Criteria:

* Adults and adolescents (age 13-75 inclusive) with a documented and confirmed pre-existing diagnosis of chronic primary immunodeficiency
* Previously or currently on IgG replacement therapy
* Documented (within 3 months) plasma IgG level of ≥500 mg/dL on current IgG therapy (IgG level can be obtained at the screening visit if documentation is not available)
* The medical records for all subjects within the previous 2 years should be available to document previous infections and treatment

Exclusion Criteria:

* Clinical evidence of any significant acute or chronic disease that, in the opinion of the investigator, may interfere with successful completion of the trial
* The subject has a known adverse reaction to Gamunex or other blood products
* The subject has a history of blistering skin disease, clinically significant thrombocytopenia, bleeding disorder, diffuse rash, recurrent skin infections or other disorders where subcutaneous therapy would be contraindicated
* The subject has known selective IgA deficiency with the exception of a known selective IgA deficient subject who has no previous documented eventful reaction to products containing IgA
* The subject is pregnant or lactating
* The subject has significant proteinuria and/or has a history of acute renal failure and/or severe renal impairment (BUN or creatinine more than 2.5 times the upper limit of normal) and/or on dialysis
* The subject has known substance or prescription drug abuse in the past 12 months
* The subject has a history of or current diagnosis of deep venous thrombosis
* The subject has an acquired medical condition that is known to cause secondary immune deficiency, such as chronic lymphocytic leukemia, lymphoma, multiple myeloma, chronic or recurrent neutropenia (absolute neutrophil count less than 1000 x 10e6/L), or HIV infection/AIDS
* The subject is receiving any of the following medications: corticosteroids (long-term daily, >1 mg of prednisone equivalent/kg/day for >30 days) (intermittent courses would not exclude subject); immunosuppressants; or immunomodulators
* The subject has non-controlled arterial hypertension (systolic blood pressure >160 mmHg and/or diastolic blood pressure >100 mmHg)
* The subject has anemia (hemoglobin <10 g/dL) at screening
* The subject has participated in another clinical trial within 30 days prior to screening (imaging studies without investigative treatments are permitted) or has received any investigational blood product within the previous 3 months

Ages: 13 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2006-11; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Sorrells, Study Director — Grifols Therapeutics LLC
Locations (8):
- United States (6):
  - University of California, Irvine, Irvine, California
  - UCLA School of Medicine, Los Angeles, California
  - Family Allergy & Asthma Center, PC, Atlanta, Georgia
  - Allergy, Asthma & Immunology Associates, PC, Omaha, Nebraska
  - Pediatric Allergy / Immunology Associates, PA, Dallas, Texas
  - Virginia Commonwealth University, Richmond, Virginia
- Canada (2):
  - Dr. Donald F. Stark, Inc, Vancouver, British Columbia
  - McGill University - Montreal General Hospital, Montreal, Quebec

REFERENCES:
- See also: FDA approved labeling information — http://www.talecris-pi.info/inserts/gamunex.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First Patient, First Visit: Nov. 21, 2006, Last patient, Last visit: Aug. 26, 2008. This study was performed at medical clinics.
Groups:
- IGIV-C: 21 subjects were required to enter a Run-In Phase (3 to 4 months) and received IGIV-C between 200 and 600 mg/kg by intravenous infusion every 3 or 4 weeks. 18 subjects completed the Run-In Phase and entered the Intravenous Phase.
  A total of 32 subjects entered the IV Phase: 14 subjects who had received IV IGIV-C prior to screening directly entered the IV Phase and 18 subjects who had completed the Run-in Phase continued in the study to enter the IV Phase. Subjects in the IV Phase received two IV infusions at the same dose (200-600 mg/kg) and frequency (every 3 or 4 weeks) as their regular dose at screening or during the Run-In Phase. All 32 subjects completed the IV Phase and entered the SC Phase.
  A total of 32 subjects who completed the IV Phase entered the SC Phase. Subjects in the SC Phase received IGIV-C via weekly SC administration for 24 weeks total at a dose that was calculated using a conversion factor and their established IV dose. 25 subjects completed the SC Phase.
Period: Run-In Phase
Arm/Group | IGIV-C
Started | 21
Completed | 18
Not Completed | 3
Not completed — Adverse Event | 1
Not completed — Lost to Follow-up | 1
Not completed — Withdrawal by Subject | 1
Period: Intravenous Phase
Arm/Group | IGIV-C
Started | 32 (18 subjects entered from the Run-in Phase and 14 new participants entered directly)
Completed | 32
Not Completed | 0
Period: Subcutaneous Phase
Arm/Group | IGIV-C
Started | 32
Completed | 25
Not Completed | 7
Not completed — Adverse Event | 2
Not completed — Non-compliance with study medication | 2
Not completed — Withdrawal by Subject | 2
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Groups:
- Safety Population: The safety population included all subjects who received any amount of study medication (IGIV-C) via intravenous (IV) and/or subcutaneous (SC) routes of administration. As such, the safety population included all study participants combined (who received any dose), whether they entered the study in the Run-In or Intravenous Phase.
Arm/Group | Safety Population
Number analyzed (Participants) | 35
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3
  Between 18 and 65 years | 28
  >=65 years | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.5 (15.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28
  Male | 7
Region of Enrollment [Number; unit: participants]
  United States | 26
  Canada | 9

OUTCOME MEASURES:

1. Primary Outcome: Geometric Least Square Means of Area Under the Curve (AUC) for Plasma Total Immunoglobulin G (IgG)
Description: Geometric least-squares mean of steady-state plasma concentration of total IgG vs. time profile (AUC).
Time Frame: IV Phase (21 or 28 days) at IV Visit #1, pre- and post-dose: 0 hr., 1 hr., and 1, 2, 3, 5, 7, 14, 21, and 28 days; SC Phase at Week #17, pre- and post-dose: 0 hr., and 1, 3, 4, 5, and 7 days
Population: A total of 32 subjects in the IV phase and 26 subjects in the SC phase had sufficient plasma concentration of total IgG vs. time profiles (AUC) for assessment of steady-state PK parameters.
Measure: Least Squares Mean (Standard Deviation); unit: mg*hr/ml
Groups:
- Gamunex Intravenous (IV) Administration: Subjects who received Gamunex via IV administration.
- Gamunex Subcutaneous (SC) Administration: Subjects who received Gamunex via SC administration.
Arm/Group | Gamunex Intravenous (IV) Administration | Gamunex Subcutaneous (SC) Administration
Number analyzed (Participants) | 32 | 26
mg*hr/ml | 7549 (1217) [0.861 to 0.917] | 6706 (1241) [0.861 to 0.917]
Statistical Analysis 1: Comparison: Gamunex Intravenous (IV) Administration vs Gamunex Subcutaneous (SC) Administration; The IV phase was considered as the Reference study phase and the SC phase as the Test study phase. The ANOVA included calculation of least-squares means (LSM), differences between adjusted means and the standard error associated with these differences; Test type: Non-Inferiority or Equivalence — The administration effect between SC and IV was assessed by exponentiation of the difference in least squares means between study phases (Test minus Reference) and the corresponding 90% confidence interval (CI) for the geometric LSM ratio between study phases (Test/Reference) for AUC. The Test (SC) was to be considered non-inferior to Reference (IV) if the lower bound of 90% CIs for the geometric LSM ratios of AUC between the Test and Reference was above 0.80 (80%); ANOVA; Geometric Least Square Mean Ratio = 0.888, 90% CI [0.861 to 0.917] — An adjusted steady-state area under the concentration vs. time curve following SC administration based on IV dosing schedule was calculated as AUC0-τ,SC multiplied by 3 or 4 for subjects on every-3-week or every-4-week IV dosing schedule

ADVERSE EVENTS:
Time Frame: Run-in phase (if required): 3 - 4 months; Intravenous Phase: 4 - 5 weeks; Subcutaneous Phase: 24 weeks.
Description: Subjects were carefully monitored for adverse events. This monitoring includes clinical and laboratory tests and physical signs such as local reactions at subcutaneous infusion sites. Adverse events were assessed in terms of their seriousness, severity, and relationship to the study drug.
Groups:
- Run-In Phase: All subjects who participated in the Run-In Phase.
- Intravenous Phase: All subjects who participated in the Intravenous Phase.
- Subcutaneous Phase: All subjects who participated in the Subcutaneous Phase.
Arm/Group | Run-In Phase | Intravenous Phase | Subcutaneous Phase
Serious Adverse Events (participants affected / at risk) | 2/21 | 0/32 | 1/32
Other Adverse Events (participants affected / at risk) | 11/21 | 9/32 | 29/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Run-In Phase (N=21) | Intravenous Phase (N=32) | Subcutaneous Phase (N=32)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sepsis syndrome (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Incisional hernia (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 0 (0)
Drug dependence (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Run-In Phase (N=21) | Intravenous Phase (N=32) | Subcutaneous Phase (N=32)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 2 (3) | 5 (8)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 4 (6)
Toothache (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 5 (6)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 2 (3)
Acute sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (5)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 3 (3)
Ear infection (Infections and infestations) | 1 (1) | 0 (0) | 2 (3)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 2 (2)
Sinusitis (Infections and infestations) | 2 (2) | 0 (0) | 8 (11)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 2 (2) | 7 (8)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 2 (2)
Viral infection (Infections and infestations) | 1 (1) | 0 (0) | 2 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 3 (6)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 2 (2)
Dizziness (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 4 (8) | 1 (1) | 6 (37)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2)
Insomnia (Psychiatric disorders) | 2 (2) | 0 (0) | 1 (1)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 3 (3)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Infusion site bruising (General disorders) | 0 (0) | 0 (0) | 7 (13)
Infusion site erythema (General disorders) | 0 (0) | 0 (0) | 13 (125)
Infusion site extravasation (General disorders) | 0 (0) | 0 (0) | 8 (13)
Infusion site haemorrhage (General disorders) | 0 (0) | 0 (0) | 5 (11)
Infusion site induration (General disorders) | 0 (0) | 0 (0) | 2 (5)
Infusion site oedema (General disorders) | 0 (0) | 0 (0) | 4 (54)
Infusion site pain (General disorders) | 0 (0) | 0 (0) | 13 (59)
Infusion site pruritus (General disorders) | 0 (0) | 0 (0) | 8 (54)
Infusion site rash (General disorders) | 0 (0) | 0 (0) | 2 (5)
Infusion site swelling (General disorders) | 0 (0) | 0 (0) | 11 (54)
Infusion site urticaria (General disorders) | 0 (0) | 0 (0) | 2 (25)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institution or Principal investigator (PI) furnishes Talecris a copy of any proposed publication (either in writing or oral) of results of the study performed under the protocol, at least 30 days before the date of submission for publication or presentation. Talecris can ask the Principal Investigator to remove Confidential Information before publication or Talecris shall have an additional time, not to exceed 60 days, to file a patent application for such Confidential Information.